CLINICAL TRIAL: NCT05661955
Title: Phase 1b/2 Study Investigating the Antitumor Activity, Safety, Tolerability, and Pharmacokinetics of the Anti-OX40 Agonist Monoclonal Antibody BGB-A445 in Combination With the Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced or Metastatic Urothelial Carcinoma, Renal Cell Carcinoma, or Melanoma
Brief Title: A Study to Investigate the Antitumor Activity, Safety, Tolerability, and Pharmacokinetics of BGB-A445 in Combination With Tislelizumab in Participants With Select Advanced Solid Tumors.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-A445-201; CTR20223270 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Urothelial Carcinoma; Renal Cell Carcinoma; Melanoma; Non-mucosal Melanoma
Keywords: Urothelial Carcinoma; Renal Cell Carcinoma; Melanoma; Advanced solid tumors; Non-mucosal melanoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Melanoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort A: Previously Treated UC (Experimental): BGB-A445 Monotherapy
  Interventions: Drug: BGB-A445
- Cohort B: Previously Treated UC (Experimental): BGB-A445 and Tislelizumab
  Interventions: Drug: BGB-A445; Drug: Tislelizumab
- Cohort C: Previously Treated RCC (Experimental): BGB-A445 Monotherapy
  Interventions: Drug: BGB-A445
- Cohort D: Previously Treated RCC (Experimental): BGB-A445 and Tislelizumab
  Interventions: Drug: BGB-A445; Drug: Tislelizumab
- Cohort E: Previously Treated Melanoma (Experimental): BGB-A445 Monotherapy
  Interventions: Drug: BGB-A445
- Cohort F: Previously Treated Melanoma (Experimental): BGB-A445 and Tislelizumab
  Interventions: Drug: BGB-A445; Drug: Tislelizumab
- Cohort G: First Line Cisplatin Ineligible UC (Experimental): BGB-A445 and Tislelizumab
  Interventions: Drug: BGB-A445; Drug: Tislelizumab
- Cohort H: First Line Non-mucosal Melanoma (Experimental): BGB-A445 and Tislelizumab
  Interventions: Drug: BGB-A445; Drug: Tislelizumab
- Cohort I: Previously Treated Non-mucosal Melanoma (Experimental): BGB-A445 and Tislelizumab
  Interventions: Drug: BGB-A445; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-A445 — administered intravenously
  Other Names: Gimistotug
Drug: Tislelizumab — administered intravenously
  Other Names: BGB-A317
  Arms: Cohort B: Previously Treated UC; Cohort D: Previously Treated RCC; Cohort F: Previously Treated Melanoma; Cohort G: First Line Cisplatin Ineligible UC; Cohort H: First Line Non-mucosal Melanoma; Cohort I: Previously Treated Non-mucosal Melanoma

SUMMARY:
The objective of this study is to assess the overall response rate, evaluate the antitumor activity, and characterize the safety and tolerability of BGB-A445 alone or in combination with tislelizumab in participants With Advanced or Metastatic Urothelial Carcinoma (UC), Renal Cell Carcinoma (RCC), or Melanoma

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants who were histologically or cytologically confirmed advanced and/or metastatic cancer. UC participants (Cohort A and B), RCC patients (Cohort C and D) or melanoma participants (Cohort E and F) who have received at least 1 but no more than 3 lines of prior systemic therapy. Cisplatin ineligible UC participants (Cohort G) who have received no prior systemic therapy and have PD-L1 CPS ≥ 10. Melanoma patients (Cohort H) with non-mucosal melanoma who have no previous systemic treatment. Melanoma participants (Cohort I) with non-mucosal melanoma who were CPI pretreated and have 1 or 2 lines of prior systemic therapy. Participants must not have received prior therapy targeting OX40 or any other T-cell agonists.
2. Has at least 1 measurable lesion as defined per RECIST v1.1.
3. Participants must be able to provide an archived formalin-fixed paraffin embedded (FFPE) tumor tissue sample
4. ECOG PS ≤ 1 (Participants with UC could have an ECOG PS ≤ 2) and a life expectancy of≥ 3 months
5. Adequate organ function as indicated by the laboratory values up to the first dose of study drug(s)

Key Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled brain metastasis
2. Active autoimmune diseases or history of autoimmune diseases that may relapse or history of life-threatening toxicity related to prior immune therapy
3. Any active malignancy ≤ 2 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent
4. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug(s), with the following exceptions:

   1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
   2. Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption
   3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a nonautoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen)
5. With uncontrolled diabetes, or > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management, or ≥ Grade 3 hypoalbuminemia occurring ≤ 14 days before the first dose of study drug(s)

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) as Assessed by the Investigator | Up to approximately 26 months
  ORR is defined as the percentage of participants who had confirmed complete response Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
Disease-Control Rate (DCR) | Up to approximately 26 months
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease as determined from tumor assessments by the investigator using RECIST v1.1.
Clinical Benefit Rate (CBR) | Up to approximately 26 months
  CBR is defined as the percentage of participants with best overall response of CR, PR, or stable disease lasting for at least 24 weeks as determined from tumor assessments by the investigator using RECIST v1.1.
Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study drugs or the initiation of new anticancer therapy, whichever comes earlier, up to 22 months
  Number of participants with AEs and SAEs characterized by type, frequency, severity (as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5.0 [NCI-CTCAE v 5.0]), timing, seriousness, and relationship to study drug(s) as needed

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (18):
- China (18):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Second Hospital and Clinical Medical School, Lanzhou University, Lanzhou, Gansu
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Jining No Peoples Hospital West Branch, Jining, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/